CLINICAL TRIAL: NCT05567367
Title: A Phase 1, Two-Part, Single-Center, Open-Label, Randomized, Cross-Over, Single Ascending Doses (SAD), Followed by a Multiple Ascending Doses (MAD) Safety and Pharmacokinetic Study of RT234 in Healthy Subjects
Brief Title: A Healthy Volunteer Study Evaluating the the Safety, Tolerability, and Pharmacokinetics of RT234
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Respira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT234-CL101; ACTRN12618001077257 (Registry Identifier: Australian New Zealand Clinical Trials Registry (ANZCTR))
Record Dates: First submitted 2022-04-04; First posted 2022-10-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer
Keywords: Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Vascular Diseases; Cardiovascular Diseases; Hypertension, Pulmonary; Lung Diseases; Respiratory Tract Diseases; Vardenafil Dihydrochloride; Inhaled Vardenafil; Vasodilator Agents; Phosphodiesterase 5 Inhibitors; Phosphodiesterase Inhibitors; Enzyme Inhibitors; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Familial Primary Pulmonary Hypertension; Vascular Diseases; Cardiovascular Diseases; Hypertension, Pulmonary; Lung Diseases; Respiratory Tract Diseases | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (6):
- RT234 0.2 mg, Single Ascending Dose (SAD) (Experimental): Part 1, SAD Cohort 1A
  Interventions: Combination Product: Drug: RT234 - vardenafil inhalation powder; Device: RS01 dry powder inhaler (RS01 DPI)
- RT234 0.6 mg followed by oral vardenafil 20mg on day 3, SAD (Experimental): Part 1, SAD Cohort 2A1
  Interventions: Combination Product: Drug: RT234 - vardenafil inhalation powder; Device: RS01 dry powder inhaler (RS01 DPI); Drug: Vardenafil Oral Tablet
- Oral vardenafil 20mg followed by RT234 0.6 mg on day 3, SAD (Experimental): Part 1, SAD Cohort 2A2
  Interventions: Combination Product: Drug: RT234 - vardenafil inhalation powder; Device: RS01 dry powder inhaler (RS01 DPI); Drug: Vardenafil Oral Tablet
- RT234 1.2 mg, SAD (Experimental): Part 1, SAD Cohort 3A
  Interventions: Combination Product: Drug: RT234 - vardenafil inhalation powder; Device: RS01 dry powder inhaler (RS01 DPI)
- RT234 2.4 mg, SAD (Experimental): Part 1, SAD Cohort 4A
  Interventions: Combination Product: Drug: RT234 - vardenafil inhalation powder; Device: RS01 dry powder inhaler (RS01 DPI)
- RT234 2.4 mg, Multiple Ascending Dose (MAD) (Experimental): Part 2, MAD Cohort 1B
  Interventions: Combination Product: Drug: RT234 - vardenafil inhalation powder; Device: RS01 dry powder inhaler (RS01 DPI)

INTERVENTIONS:
Combination Product: Drug: RT234 - vardenafil inhalation powder; Device: RS01 dry powder inhaler (RS01 DPI) — RT234 is a drug/device combination product composed of vardenafil hydrochloride as the drug constituent and will utilize RS01 DPI device.
  Other Names: vardenafil inhalation powder
Drug: Vardenafil Oral Tablet — 20 mg oral vardenafil tablet.
  Other Names: Levitra
  Arms: Oral vardenafil 20mg followed by RT234 0.6 mg on day 3, SAD; RT234 0.6 mg followed by oral vardenafil 20mg on day 3, SAD

SUMMARY:
The objective of this two part study was to demonstrate safety, tolerability, and pharmacokinetics of RT234 in healthy volunteers.

This study is also known as Vardenafil Inhaled for Pulmonary Arterial Hypertension PRN Phase 1 (VIPAH-PRN 1) study

DETAILED DESCRIPTION:
This study was designed to evaluate safety and tolerability and to characterize the PK profiles of single and repeated doses of inhaled vardenafil as RT234. In addition, vardenafil PK after single 0.6 mg doses of RT234 was compared to that following administration of a single 20 mg dose of oral vardenafil tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female, 18 to 45 years of age (inclusive at time of informed consent)
2. Normal heart, lung, kidney, and liver function based on physical examination
3. Systolic blood pressure of 100-145 mmHg, diastolic blood pressure of 50-90 mmHg, and a resting heart rate of 40-100 bpm at Screening
4. A body mass index (BMI) of ≤18 to ≥30 kg/m2 at Screening
5. Must be a non-smoker or ex-smoker with less than a 5-pack year history of smoking (including the use of electronic cigarettes) and have ceased smoking ≥1 year prior to Screening; or a social smoker (defined as less than 10 cigarettes in the previous 12 months)

Exclusion Criteria:

1. Has serum transaminase (i.e., alanine aminotransferase [ALT], aspartate aminotransferase [AST], or gamma-glutamyl transferase [GGT]) levels greater than three times the upper level of normal
2. Abnormal orthostatic vital signs (at screening) defined as a decrease of ≥20 mmHg in systolic blood pressure and/or a decrease of ≥10 mmHg in diastolic blood pressure and/or >25 bpm increase in heart rate within 3 minutes of standing, or with symptoms of light-headedness, dizziness, or fainting upon standing.
3. History of hypotension including fainting, syncope, orthostatic hypotension, and/or vasovagal reactions
4. History of retinitis pigmentosa
5. Vision loss due to non-arteritic anterior ischemic optic neuropathy (NAION) or other optic perfusion impairment
6. History of priapism or anatomical deformation of the penis
7. History of sudden sensorineural hearing loss (SSHL), need for hearing aids, and/or other documented hearing loss
8. A corrected QT interval using Fridericia's formula (QTcF) >450 msec
9. Has evidence of significant obstructive lung disease on spirometry. Subjects with any of the following criteria will be excluded:

   1. FEV1 <60% (predicted) (pre-bronchodilators); or
   2. FEV1/FVC <65% (pre-bronchodilators)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment related adverse events as assessed by CTCAE v5.0 | Up to to 10 days
  Adverse events reported by participants and those observed by the investigator in relation to laboratory tests, vital signs, ECGs, medications used to treat adverse events, and physical examinations were analyzed.

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | Up to 10 days
  Cmax was measured for 4 single doses of oral vardenafil.
Time to reach maximum concentration (Tmax) | Up to 10 days
  Tmax was measured for 4 single doses of oral vardenafil.
Area under the curve (AUC) | Up to 10 days
  AUC was measured for 4 single doses of RT234
Half life (t1/2) | Up to 10 days
  t1/2 was measured for 4 single doses of RT234
Terminal elimination rate constant (Kel) | Up to 10 days
  Kel was measured for 4 single doses of RT234
Total body clearance (CL/F) | Up to 10 days
  CL/F was measured for 4 single doses of RT234
Total volume of distribution at the terminal phase | Up to 10 days
  measured for 4 single doses of RT234

CONTACTS AND LOCATIONS:
Overall Officials: Donna Jarlenski, MS, Study Director — Respira Therapeutics
Locations (1):
- Nucleus Network, Burnet Institute, Prahran, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eldon MA, Parsley EL, Maurer M, Tarara TE, Okikawa J, Weers JG. Safety, Tolerability, and Pharmacokinetics of RT234 (Vardenafil Inhalation Powder): A First-in-Human, Ascending Single- and Multiple-Dose Study in Healthy Subjects. J Aerosol Med Pulm Drug Deliv. 2021 Aug;34(4):251-261. doi: 10.1089/jamp.2020.1651. Epub 2020 Dec 15. PMID 33325799